CLINICAL TRIAL: NCT04118361
Title: Eye-ECG Approach to Emergencies : Diagnostic Performance of the HINTS Test Performed by Emergency Physicians to Distinguish a Central Cause From a Peripheral Cause of Isolated Acute Vestibular Syndrome
Brief Title: Eye-ECG Approach to Emergencies : Diagnostic Performance of the HINTS Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Eye-ECG approach
Record Dates: First submitted 2019-09-23; First posted 2019-10-08 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Acute Vestibular Syndrome; Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with AVS isolated at emergencies (Experimental): Enrollment of patients with AVS isolated at emergencies
  Interventions: Diagnostic Test: HINTS Test; Diagnostic Test: STANDING Algorithm

INTERVENTIONS:
Diagnostic Test: HINTS Test — The HINTS test is a clinical test composed of 3 oculomotor examinations:
  * Search for high-frequency vestibulo-ocular reflex during a passive head impulse test
  * Highlighting of spontaneous nystagmus: it must be sought without, then with Frenzel glasses because they allow to temporarily interrupt the ocular fixation.
  * Vertical divergence
  This test is performed at the patient's bedside in about 3 minutes. Presence of at least one of the three items of central locator value is sufficient to diagnose a central cause of VAS, including normal early brain imaging.
Diagnostic Test: STANDING Algorithm — The STANDING algorithm consists of clinical elements that can be evaluated in about 10 minutes at the patient's bedside: two oculomotor examinations (Head Impulse Test and detection of a nystagmus), detection of ataxia and the practice of release maneuvers.

SUMMARY:
Vertigo integrated with acute vestibular syndrome (AVS) is a frequent reason for emergency visits. The French and international literature estimates between 2 to 4% of vertigo prevalence among reasons for coming to emergencies. International classifications define AVS as vertigo or acute dizziness (less than one month) and persistent, gait instability, nausea or vomiting, nystagmus or an intolerance to head movements.

In emergency departments, the clinical approach of vertiginous patients is difficult because the "vertigo" term is sometimes used in by patients, or because they use the terms "uneasiness", "vertigo", or "dizziness" without distinction. These terms sometimes include various sensations of "sleeping head", "blurred vision", "instability", "pitch" etc. A first difficulty is therefore to clarify these terms and organize syndrome expressed by the patient. A rigorous interrogation is therefore essential and can be time-consuming.

Another difficulty is to carry out an exhaustive clinical examination including the assessment of the general condition and hydration, an ENT examination and a neurological examination. However, at the end of these steps, the orientation central or peripheral etiology is not simple. In the last consensus conference of the Barany Society (2014) the classification of VAS into three types was not sufficient to distinguish "benign" vertigo from "risky" dizziness (related to a central cause).

DETAILED DESCRIPTION:
The HINTS test (Head Impulse, Nystagmus, Test of Skew) is a clinical test composed of 3 oculomotor examinations: the search for high frequency vestibulo-ocular reflex during a passive impulse of the head (Head Impulse test), the detection of a spontaneous nystagmus and a vertical divergence. It has been developed to evaluate patients with AVS defined as vertigo or acute and persistent dizziness sometimes accompanied by nausea or vomiting, and/or gait instability, and/or nystagmus, and/or intolerance to head movements. This time saving is important, as a complete neurological examination usually takes between 10 and 15 minutes. The presence of at least one of the three items of central locator value is sufficient to diagnose a central cause of AVS, including normal early brain imaging. Some studies suggest that absence of these three criteria does not require an emergency neuroimaging examination and allows ambulatory management of the patient, in search of a peripheral cause of the ENT sphere.

The STANDING clinical algorithm (SponTAneous, Nystagmus, Direction, head Impulse test, STANDING) was proposed by Vanni in 2015 for diagnosis of the AVS central causes in emergencies in a one-year prospective Italian monocentric study. The STANDING algorithm consists of clinical elements that can be evaluated in about 10 minutes at the patient's bedside: two oculomotor examinations (Head Impulse Test and detection of a nystagmus), detection of ataxia and practice of release maneuvers.

Currently, the patient management with isolated AVS in the emergency room lacks an ideal diagnostic clinical test: efficient, non-invasive, inexpensive and painless.

The investigators would like to know what diagnostic performance of the HINTS test (sensitivity and specificity) is when it is performed by emergency physicians on a population of patients with isolated AVS in emergency room. They can thus either be part of non-urgent outpatient care in the event of suspicion of a peripheral cause of the ENT sphere, or part of rapid and aggressive inpatient neurological care in the event of suspicion of a central cerebral cause.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking patient.
* Affiliated with social security or, failing that, with another health insurance system.
* Patient capable of giving free, informed and express consent
* Patient with an isolated AVS defined by a progression of more than one hour and less than one month and at least one of the following criteria:
* Vertigo (illusion of the subject moving in relation to surrounding objects or objects) surrounding with respect to the subject, a sensation of rotation, movement of the body in the plane vertical, unstable, described as a pitch or "rotating head"), sometimes associated with vegetative signs (nausea, vomiting, pallor, sweating, slowing of frequency cardiac),
* A nystagmus (spontaneous or positional),
* Ataxia characterized by gait disorders with imbalance type (which can dominate the symptomatology) with sways, a brittle gait or simple instability.

A patient may be included several times during the study period provided that they are acute episodes separate.

Exclusion Criteria:

* Patient with focal neurological signs concomitantly appearing with AVS: disorder of the language or writing, speech impairment, dysarthria, movement performance disorders voluntary, sensory motor deficit, involuntary abnormal movements. The vertiginous patients with ataxia meet the inclusion criteria provided they do not show any other sign neurological focal, in particular, other signs of cerebellar syndrome.
* Patient with a Glasgow score <15 or blood glucose < 0.70 g/l, MAP < 65 mm Hg, acute anemia and <7g/dl, transient dizziness having disappeared upon arrival in the emergency room, acute alcohol abuse, acute alcohol abuse, and acute drug intoxication, a history of oculomotor paralysis.
* Patient under guardianship or curatorship.
* Patient deprived of liberty.
* Patient under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of the HINTS test performed by pre-trained emergency doctors (DEMs) to distinguish a central cause from a peripheral cause in a patient with isolated VAS in the emergency department | Day 1
  This outcome measure the sensitivity of the HINTS test performed by a DEM in emergencies for the diagnosis of central and peripheral causes.
Diagnostic specificity of the HINTS test performed by pre-trained emergency doctors (DEMs) to distinguish a central cause from a peripheral cause in a patient with isolated VAS in the emergency department | Day 1
  This outcome measure the specificity of the HINTS test performed by a DEM in emergencies for the diagnosis of central and peripheral causes.

SECONDARY OUTCOMES:
Diagnostic sensitivity of the STANDING algorithm performed by DEMs to distinguish a cause of a peripheral cause in a patient with isolated AVS in the emergency department; then compare this performance to the HINTS test | Day 1
  This Outcome measure the sensitivity by the STANDING algorithm performed by a DEM in emergencies for the diagnosis of central and peripheral causes.
  - Performance difference between the HINTS test and the STANDING algorithm
Diagnostic specificity of the STANDING algorithm performed by DEMs to distinguish a cause of a peripheral cause in a patient with isolated AVS in the emergency department; then compare this performance to the HINTS test | Day 1
  This Outcome measure the specificity by the STANDING algorithm performed by a DEM in emergencies for the diagnosis of central and peripheral causes.
  - Performance difference between the HINTS test and the STANDING algorithm
Opinion of trained doctors on the use and interpretation of the HINTS test and STANDING algorithm | Day 1
  This outcome is to answer the opinion of trained doctors on the use and interpretation of the HINTS test and the STANDING algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Camille GERLIER, M.D, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Tarnutzer AA, Berkowitz AL, Robinson KA, Hsieh YH, Newman-Toker DE. Does my dizzy patient have a stroke? A systematic review of bedside diagnosis in acute vestibular syndrome. CMAJ. 2011 Jun 14;183(9):E571-92. doi: 10.1503/cmaj.100174. Epub 2011 May 16. No abstract available. PMID 21576300
- [Background] Kerber KA, Meurer WJ, Brown DL, Burke JF, Hofer TP, Tsodikov A, Hoeffner EG, Fendrick AM, Adelman EE, Morgenstern LB. Stroke risk stratification in acute dizziness presentations: A prospective imaging-based study. Neurology. 2015 Nov 24;85(21):1869-78. doi: 10.1212/WNL.0000000000002141. Epub 2015 Oct 28. PMID 26511453
- [Background] Kene MV, Ballard DW, Vinson DR, Rauchwerger AS, Iskin HR, Kim AS. Emergency Physician Attitudes, Preferences, and Risk Tolerance for Stroke as a Potential Cause of Dizziness Symptoms. West J Emerg Med. 2015 Sep;16(5):768-76. doi: 10.5811/westjem.2015.7.26158. Epub 2015 Oct 20. PMID 26587108
- [Background] Kattah JC, Talkad AV, Wang DZ, Hsieh YH, Newman-Toker DE. HINTS to diagnose stroke in the acute vestibular syndrome: three-step bedside oculomotor examination more sensitive than early MRI diffusion-weighted imaging. Stroke. 2009 Nov;40(11):3504-10. doi: 10.1161/STROKEAHA.109.551234. Epub 2009 Sep 17. PMID 19762709
- [Background] Newman-Toker DE, Kerber KA, Hsieh YH, Pula JH, Omron R, Saber Tehrani AS, Mantokoudis G, Hanley DF, Zee DS, Kattah JC. HINTS outperforms ABCD2 to screen for stroke in acute continuous vertigo and dizziness. Acad Emerg Med. 2013 Oct;20(10):986-96. doi: 10.1111/acem.12223. PMID 24127701
- [Background] Becares-Martinez C, Lopez-Llames A, Arroyo-Domingo MM, Marco-Algarra J, Morales Suarez-Varela MM. [What do MRI and CT scan provide us in patients with vertigo and dizziness? A cost-utility analysis]. Rev Neurol. 2019 Apr 16;68(8):326-332. doi: 10.33588/rn.6808.2018399. Spanish. PMID 30963529
- [Background] Dumitrascu OM, Torbati S, Tighiouart M, Newman-Toker DE, Song SS. Pitfalls and Rewards for Implementing Ocular Motor Testing in Acute Vestibular Syndrome: A Pilot Project. Neurologist. 2017 Mar;22(2):44-47. doi: 10.1097/NRL.0000000000000106. PMID 28248913
- [Background] Vanni S, Nazerian P, Casati C, Moroni F, Risso M, Ottaviani M, Pecci R, Pepe G, Vannucchi P, Grifoni S. Can emergency physicians accurately and reliably assess acute vertigo in the emergency department? Emerg Med Australas. 2015 Apr;27(2):126-31. doi: 10.1111/1742-6723.12372. Epub 2015 Mar 10. PMID 25756710
- [Result] Gerlier C, Hoarau M, Fels A, Vitaux H, Mousset C, Farhat W, Firmin M, Pouyet V, Paoli A, Chatellier G, Ganansia O. Differentiating central from peripheral causes of acute vertigo in an emergency setting with the HINTS, STANDING, and ABCD2 tests: A diagnostic cohort study. Acad Emerg Med. 2021 Dec;28(12):1368-1378. doi: 10.1111/acem.14337. Epub 2021 Jul 20. PMID 34245635